CLINICAL TRIAL: NCT02333305
Title: Evolution of Albumin on AOA1 Patients Supplemented With Coenzyme Q10
Acronym: AOA1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P081107
Record Dates: First submitted 2014-09-29; First posted 2015-01-07 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Ataxia-oculomotor Apraxia 1
Keywords: Ataxia with Oculomotor Apraxia type 1; CoQ10; hypoalbuminemia
MeSH Terms: conditions — Early-onset ataxia with oculomotor apraxia and hypoalbuminemia; Hypoalbuminemia | interventions — coenzyme Q10

STUDY DESIGN:
Intervention Model Description: coenzyme Q10
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Coenzyme Q10 (CoQ10) - is a Dietary complement that contains Coenzyme Q10 (Ubidecarenone) well characterized nano particles.
  Interventions: Dietary Supplement: CoQ10
- 2 (Placebo Comparator): Placebo of CoQ10 is a translucent nano-emulsion of well characterized nano particles. Lecithin (and) Alcohol (and) Glycerin (and) Aqua
  Interventions: Other: Sanomit Placebo

INTERVENTIONS:
Dietary Supplement: CoQ10 — • 2 dosages according to patient weight: Weight < 50kg : 20 drops 3 times a day (150 mg / d) Weight ≥ 50 kg : 40 drops 3 times a day (300 mg / d)
  Arms: 1
Other: Sanomit Placebo — • according to patient weight: Weight < 50kg : 20 drops 3 times a day Weight ≥ 50 kg : 40 drops 3 times a day
  Arms: 2

SUMMARY:
We propose a study on Ataxia with oculomotor apraxia type 1 (AOA1) in which Coenzyme Q10 (CoQ10) deficit has been observed. Main objectives of the study are :

* To monitor evolution of albumin in patients affected with AOA1 while supplemented with CoQ10 ;
* To measure with clinical scales and biological markers efficacy of supplementation on disease evolution.

AOA1 is characterised by Hypoalbuminemia. Disease duration is negatively correlated with albumin level. This study aims to understand mechanisms of the disease and our hypothesis is that correction or stabilization of albumin level with CoQ10 supplementation could impact disease evolution. The study is planned from 1 to 2 years supplementation. The CoQ10 is classified as a food supplement and has already been tested in other neurological conditions.

DETAILED DESCRIPTION:
Ataxia with ocular apraxia type 1 (AOA1) is an autosomal recessive cerebellar ataxia. Patients' phenotype associates early onset cerebellar ataxia, oculomotor apraxia, neuropathy and often intellectual disability, hypoalbuminaemia and hypercholesterolemia.

APTX gene mutations responsible for AOA1 disease were identified in a family previously reported with ataxia and Coenzyme Q10 deficiency. Therefore we measured muscle Coenzyme Q10 in six patients AOA1 and found decreased levels in five. Hypercholesterolaemia and low albumin levels represent hallmarks of the disease.

We thus propose therapeutic trial with Coenzyme Q10 in AOA1 patients, by using albumin evolution as primary endpoint.

Moreover several secondary endpoints will be performed:

* clinical examination (SARA scale)
* quantitative assessments of the ataxia (with the calculation of the Composite Cerebellar Functional Severity CCFS)
* biological criteria (prealbumin, cholesterol, alphafoetoprotein, blood count, hepatic checkup)
* oculographic examination.

The study is a multicentric randomised placebo controlled trial with two-year follow-up:

* during the first year, one group will be supplemented with Coenzyme Q10 while the other group will receive a placebo;
* during the second year, all patients will be supplemented with Coenzyme Q10 in order to assess long term safety and tolerance of the treatment.

ELIGIBILITY:
Inclusion criteria :

* 1. Diagnosis of ataxia with oculomotor apraxia type I (AOA1) confirmed by genetic molecular analysis
* 2. Age ≥ 18 years
* 3. Hypoalbuminemia
* 4. Efficient contraception for women of childbearing potential (with pregnancy test during each visit)
* 5. Signature of the written informed consent form
* 6. Presence of a support person (for patient with cognitive disorders)

Exclusion criteria :

* 1. Hypersensitivity to one of the excipients (glycerin, ethanol, lecithin)
* 2. Absence of hypoalbuminemia
* 3. During the 2 months before inclusion :

  * Use of CoQ10
  * Treatment with antioxidants (vitamin C) and statins
  * Use of drugs affecting mitochondrial activity
  * Anti-cholesterol, thyroid hormones, anti-arrhythmic compounds, warfarin, metformin or clozapine
* 4. Treatment with vitamin E, calcium, magnesium and/or other vitamins with a concentration superior to 149 UI during more than 3 months before inclusion
* 5. Use of drugs interfering with catacholamine metabolism (reserpine, amphetamine, or inhibitors of the monoamine oxidase A, methylphenidate, cinnarizine) during the month before inclusion
* 6. Non balanced treatment with anxiolytics, hypnotics, tranquillizers and/or antidepressants during the month before inclusion
* 7. Hypothyroidism with thyroxin use
* 8. Epilepsy
* 9. Psychotic disorders
* 10. Pregnancy or lactation period
* 11. Woman of childbearing potential without efficient contraception
* 12. Participant to other therapeutic studies during the month before inclusion
* 13. Inability to receive a clear information on the research
* 14. Inability to participate to the totality of the study
* 15. Non affiliation to social security (beneficiary or assignee)
* 16. Refusal of signing the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-06; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Albuminemia | 2 years
  Evolution of albuminemia every 6 months during 2 years.

SECONDARY OUTCOMES:
SARA scale | 2 years
  Evolution of clinical criteria (SARA and CCFS, which represent quantitative scales to assess cerebellar ataxia evolution)
CCFS | 2 years
  Evolution of clinical criteria (SARA and CCFS, which represent quantitative scales to assess cerebellar ataxia evolution)
prealbuminemia | 2 years
  Evolution of biological criteria (prealbuminemia, cholesterol, alfa-foeto-protein) every 6 months during 2 years.
cholesterol | 2 years.
  Evolution of biological criteria (prealbuminemia, cholesterol, alfa-foeto-protein) every 6 months during 2 years.
alfa-foeto-protein | 2 years.
  Evolution of biological criteria (prealbuminemia, cholesterol, alfa-foeto-protein) every 6 months during 2 years.
Oculomotor evaluation | 2 years
  Oculomotor evaluation to assess oculo motor apraxia evolution [Time Frame: Each year during 2 years.]
EQ5D - PHQ9 | 2 years
  Quality of life evolution (self-administered questionnaire EQ5D - PHQ9) every 6 months during 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Perrine Charles, MD, PhD, Principal Investigator — Assitance Publique - Hopitaux de Paris
Locations (1):
- ICM Institute, Paris, France

IPD SHARING:
Plan to Share IPD: No